CLINICAL TRIAL: NCT06698991
Title: Daily Versus Alternate Day Plasma Exchange in Wilson Disease With Acute Liver Failure in Children: A Randomized Controlled Trial
Brief Title: Daily Versus Alternate Day Plasma Exchange in Wilson Disease With Acute Liver Failure in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALF-07
Record Dates: First submitted 2024-11-16; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Acute Liver Failure; Wilson Disease
MeSH Terms: conditions — Liver Failure, Acute; Hepatolenticular Degeneration | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily plasma exchange + SMT (Experimental): (Maximum 3+1 sessions during a period of 7 days)
  Interventions: Biological: Plasma Exchange; Other: Standard Medical Treatment
- Alternate day therapeutic plasma exchange + SMT (Active Comparator): Alternate day therapeutic plasma exchange + SMT
  Interventions: Biological: Plasma Exchange; Other: Standard Medical Treatment

INTERVENTIONS:
Biological: Plasma Exchange — • Plasma exchange (1.5 times plasma exchange)
  * Blood volume: 80ml/kg
  * Plasma volume = Blood volume x (1 - Hematocrit/100)
  * TPE volume = 1.5 x plasma volume
  * Duration: 4 hours
Other: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
Wilson disease in children has a varied presentation. Wilson disease with acute liver failure is associated with very high mortality and morbidity. The standard therapy i.e chelation (with either D- penicillamine or trientene can be used as a temporizing agent to treat the enormous release of copper into the blood stream; however, substantial removal is not achieved for at least 1 to 3 months. Plasma exchange provides a means of rapid means of removal of copper. As per American Society for Apheresis, TPE in wilson disease with acute liver failure can rapidly remove an average of 20 mg of copper per TPE treatment. Decreased serum copper may decrease hemolysis, prevent progression of kidney failure and provide clinical stabilization. TPE can also remove large molecular weight toxins (aromatic amino acids, ammonia, endotoxins) and other factors, which may be responsible for hepatic coma. The frequency of said TPE is not defined as most evidence is based on case reports and case series.

Copper is highly protein bound and the volume of distribution for copper is large. Under normal conditions, 90-95% of serum copper is ceruloplasmin-bound with the remaining 5-10% being nonceruloplasmin-bound. TPE efficiently removes both ceruloplasmin- and albumin-bound copper. FFP used for exchange can be helpful in treating the associated coagulopathy. TPE has been used as a bridge to liver transplantation as well as seen to improve survival with native liver, the optimum protocol for same remains uncertain.

DETAILED DESCRIPTION:
Study population: Children aged 3 to 18 years with Wilson disease (diagnosed as per Leipzig score >=4) with fulminant presentation (as defined by New Wilson Index>= 11 and INR >= 2.5 ).

Adverse effects: Therapeutic plasma exchange has been shown to be safe and effective in improving native liver survival in Wilson disease patients and is currently standard of care in patients with wilson disease with acute liver failure. However, TPE can be associated with risk of adverse events like infections, fluid overload or circulatory insufficiency, hypersensitivity to blood products.

Stopping rule:

1. Septic Shock
2. Anaphylaxis to blood products
3. HE grade3/4
4. INR > 5 any time point
5. INR >3.5 24 hours after 3 HVP Patients fulfilling criteria 3, 4 and 5 would be listed for liver transplantation. In case of 1, 2 appropriate medical management will be done as per department protocol.

Intervention:

Group 1: Daily plasma exchange + SMT (Maximum 3+1 sessions during a period of 7 days) Group 2: Alternate day therapeutic plasma exchange + SMT

ELIGIBILITY:
Inclusion Criteria:

1. Wilson disease with New Wilson Index of ≥ 11 and INR ≥ 2.5
2. Children aged 3 years to 18 years

Exclusion Criteria:

1. Grade 3 or grade 4 hepatic encephalopathy
2. Septic shock
3. Disseminated intravascular coagulation
4. Marked hemodynamic instability requiring a high dose of vasopressors (norepinephrine >0.5 mcg/kg/min)
5. Any severe cardio-pulmonary pre-existing disease

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the reduction in NWI (New Wilson Index) between both groups at the end of three sessions of plasma exchange | 7 days
  The New Wilson Index is a composite score containing of bilirubin, albumin, INR, AST, total leucocyte count ranging from minimum score of 0 till maximum of 20 with a higher score correlating with a worse outcome. A score of NWI >=11 is associated with increased mortality and considered an indication for consideration for liver transplantation in patients with Wilson disease.

SECONDARY OUTCOMES:
Comparison of change in serum and urine copper levels on day 7 after initiation of plasmapheresis as compared to baseline in alternate versus daily plasma exchange group. | Day 7
Comparison of overall and native liver survival at day 90 between the two groups | 90 days
Comparison of change in dialysate copper levels at the end of 3rd session between both groups. | 1 week
Comparison of total number of sessions of plasma exchange between both groups as on day 28. | Day 28
Comparison of AST in U/L, ALT in U/L at end of 3rd plasma exchange compared to baseline. | 1 week
Comparison of corrected reticulocyte count (percentage) at end of 3rd plasma exchange compared to baseline. | 1 week
Comparison of International Normalised Ratio (INR) at end of 3rd plasma exchange compared to baseline. | 1 week
Comparison of bilirubin (mg/dL) at end of 3rd plasma exchange compared to baseline. | 1 week
Comparison of albumin (mg/dL) at end of 3rd plasma exchange compared to baseline. | 1 week
Comparison of serious adverse events as defined by CTCAE criteria in both the groups. | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided